CLINICAL TRIAL: NCT00470145
Title: A Randomised, Single Blind, 2 Period, Crossover Study to Compare the Single Dose Pharmacokinetics and Tolerability of Formulations Containing Unmilled and Micronised SB-568859 in Healthy Adults
Brief Title: Comparison Of Two Tablet Formulations Of SB-568859
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: LP4110001
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-02

CONDITIONS: Atherosclerosis
Keywords: unmilled formulation,; micronised formulation; relative bioavailability,
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SB-568859

SUMMARY:
SB-568859 is a medication that is being developed for the treatment of atherosclerosis (hardening of the arteries). The purpose of this study is to see if there is a difference in how the human body takes up the study drug depending on how the study drug is made. This study will compare SB-568859 tablets that are made in 2 different ways. This is not a treatment study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and sterile women between 18 and 50 years old
* Body weight greater than 50 pounds and a body mass index between 19 and 31
* Normal electrocardiogram

Exclusion criteria:

* No history of asthma or severe allergic reactions
* No history of or current drug use
* No Hepatitis or HIV/AIDS
* No excessive alcohol use
* No smoking or tobacco use
* No use of prescription drugs, over-the-counter drugs or vitamins within 7 days
* No use of herbal supplements within 14 days
* No treatment with an investigational drug within 30 days.
* No treatment with 4 or more investigational drugs in the last 12 months
* No grapefruit or grapefruit juice in the last 7 days
* No donation of blood in the last 8 weeks
* No history of allergy to heparin
* No history of liver or gall bladder disease
* Unwillingness to use contraception

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2007-04; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Comparison of the amount of SB-568859 found in the blood over a period of 6 days after a single dose of each of the two types of tablets | 6 days

SECONDARY OUTCOMES:
Assessment of the safety and tolerability of SB-568859 after a single dose of each of the two types of tablets based on blood and urine tests, vital signs, electrocardiograms and reporting of side effects over a period of 6 days after each dose. | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States